CLINICAL TRIAL: NCT04379700
Title: Feasibility and Safety of Geniculate Artery Embolization for Treatment of Mild to Moderate Knee Osteoarthritis
Brief Title: Geniculate Artery Embolization for Treatment of Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-00370
Record Dates: First submitted 2020-05-06; First posted 2020-05-07 (Actual); Results first posted 2025-05-31 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Embolization Group (Experimental): 23 participants who are aged between 30 to 75 years old, with grade 2 or 3 knee OA on the most recent knee radiographs obtained within 6 months of intervention. Each individual participant will be enrolled for approximately 13 months to complete all study visits from the initial screening visit to last follow up at 12-months post intervention.
  Interventions: Procedure: Transcatheter arterial embolization; Device: Embozene™ Microspheres

INTERVENTIONS:
Procedure: Transcatheter arterial embolization — Transcatheter arterial embolization of one or more genicular artery(ies) using Embozene™ Color-Advanced Microspheres. Embozene™ Color-Advanced Microspheres are spherical, tightly calibrated, biocompatible, non-resorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer used for embolization.
Device: Embozene™ Microspheres — Embozene™ Microspheres are spherical, tightly calibrated, biocompatible, nonresorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer (Polyzene™-F). The microspheres intended to occlude vasculature for the purpose of blocking blood flow to a target tissue. They are available in prefilled syringes in a range of sizes suitable for embolic therapy. The microspheres are compressible to enable smooth delivery through the indicated delivery catheter and color-coded by size to allow for easy identification. 250 μm microsphere will be used and are supplied in prefilled yellow syringes.

SUMMARY:
Single-arm, single-center, no sham or placebo, prospective pilot trial designed to evaluate the feasibility and safety of transcatheter arterial embolization in patients with mild to moderate radiographic knee OA. Eligible participants will receive geniculate artery embolization using Embozene™ Color-Advanced Microspheres. Patients will be followed up for a total of 12 months.

DETAILED DESCRIPTION:
The current study seeks to determine whether transcatheter arterial embolization of abnormal neovasculature arising from the genicular arterial branches is safe and effective in the treatment of mild-to-moderate knee OA.

ELIGIBILITY:
Inclusion Criteria:

1. 30-80 years of age of any gender;
2. Kellgren-Lawrence Grade 2, 3, or 4 (in select subjects who have no bony deformity) knee OA on most recent knee radiograph obtained within 6 months of screening visit;
3. Knee pain resistant to conservative treatment for at least 3 months (anti- inflammatory drugs, acetaminophen, physical therapy, muscle strengthening, or intra- articular injection of hyaluronic acid and/or steroids);
4. Moderate to severe knee pain: pain VAS ≥ 40 mm with 0 representing 'no pain' and 100 'the worst pain imaginable. If both knees meet inclusion criteria, the one with a higher VAS score will be chosen for the study (i.e., target knee).
5. Willing, able, and mentally competent to provide informed consent and complete study questionnaires in English. The Study questionnaire is validated in English.

Exclusion Criteria:

1. Active systemic or local knee infection;
2. Active malignancy;
3. Life expectancy less than 12 months;
4. Prior ipsilateral knee surgery (within 3 years of baseline visit), arthroscopic surgery (within 6 months of baseline), total or partial knee replacement regardless of timing;
5. Ipsilateral knee intra-articular injection in the last 3 months;
6. Rheumatoid arthritis, spondyloarthropathies, crystal disease, gout, pseudogout, or lupus;
7. Pregnant during the study period;
8. Renal dysfunction as defined by serum creatinine >1.6 dl/mg or eGFR <60 on blood tests obtained within 30 days of procedure;
9. Body weight greater than 200 Kg;
10. Uncorrectable coagulopathy (platelet count < 50,000, international normalized ratio >1.5 within 30 days of procedure;
11. Known history of contrast allergy resulting in anaphylaxis;
12. Known significant arterial atherosclerosis that would limit selective angiography and/or lower extremity symptoms thought to be secondary to arterial vascular disease (eg claudication, ischemic rest pain);
13. Post-traumatic knee (if trauma occurred within 12 months of baseline or was associated with fractures);
14. Known avascular necrosis in the target knee;
15. Contraindications to MRI such as such as claustrophobia, metallic fragment/implants, pacemaker.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-03-12 (Actual); Study Completion 2025-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bedros Taslakian, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a small scale, single-site research study for NYU

RESULTS

PARTICIPANT FLOW:
Groups:
- Embolization Group: Participants who are aged between 30 to 75 years old, with grade 2 or 3 knee OA on the most recent knee radiographs obtained within 6 months of intervention. Each individual participant will be enrolled for approximately 13 months to complete all study visits from the initial screening visit to last follow up at 12-months post intervention.
  Transcatheter arterial embolization: Transcatheter arterial embolization of one or more genicular artery(ies) using Embozene™ Color-Advanced Microspheres. Embozene™ Color-Advanced Microspheres are spherical, tightly calibrated, biocompatible, non-resorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer used for embolization.
  Embozene™ Microspheres: Embozene™ Microspheres are spherical, tightly calibrated, biocompatible, nonresorbable, hydrogel microspheres coated with an inorganic perfluorinated polymer (Polyzene™-F). The microspheres intended to occlude vasculature for the purpose of blocking blood flow to a target tissue. They are available in prefilled syringes in a range of sizes suitable for embolic therapy. The microspheres are compressible to enable smooth delivery through the indicated delivery catheter and color-coded by size to allow for easy identification. 250 μm microsphere will be used and are supplied in prefilled yellow syringes.
Period: Overall Study
Arm/Group | Embolization Group
Started | 38
Participants Received GAE Treatment | 25
Completed | 21
Not Completed | 17
Not completed — Withdrawal by Subject | 10
Not completed — Screen Fail | 4
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 19
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 17
  More than one race | 0
  Unknown or Not Reported | 5
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) - Pain Score
Description: The WOMAC questionnaire includes 24 questions on daily activities. The Pain Score subsection includes five questions regarding pain (pain during walking, stair climbing, nocturnal, rest, weight bearing); each question is scored on a Likert scale as follow: 0 for no pain, 1 for mild, 2 for moderate, 3 for severe, and 4 for extreme pain. The total score is the sum of responses and ranges from 0-20; higher scores indicate greater pain.
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 24
Percentage change | -50.1 (26.4)

2. Secondary Outcome: Change in WOMAC - Pain Score
Description: as for outcome 1
Time Frame: Baseline, Month 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Percentage change | -39.6 (36.7)

3. Secondary Outcome: Change in WOMAC - Pain Score
Description: as for outcome 1
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 21
Percentage change | -43.70 (48.9)

4. Secondary Outcome: Change in Visual Analogue Scale (VAS) Rating of Knee Pain
Description: The electronic VAS is a horizontal line with no markings on the scale except "No pain" on the left (score: 0 mm) and "worst possible pain" on the right end of the scale (score: 100 mm). Subjects mark the VAS to indicate their current pain level, with 0 mm representing "No pain" and 100 mm representing "worst possible pain".
Time Frame: Baseline, Month 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Percentage change | -48.50 (33.6)

5. Secondary Outcome: Change in VAS Rating of Knee Pain
Description: as for outcome 4
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 24
Percentage change | -50.80 (37.9)

6. Secondary Outcome: Change in VAS Rating of Knee Pain
Description: as for outcome 4
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 21
Percentage change | -55.40 (3770.00)

7. Secondary Outcome: Change in WOMAC - Stiffness Score
Description: The WOMAC - Stiffness Score is calculated using the Knee Injury and Osteoarthritis Outcome Score (KOOS) extension to the WOMAC score. The Stiffness Score comprises 2 items related to knee stiffness; both items are rated on a Likert scale from 0-4; the total score is the sum of responses and ranges from 0-8. Higher scores indicate more severe knee stiffness.
Time Frame: Baseline, Month 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Percentage change | -39.80 (41.5)

8. Secondary Outcome: Change in WOMAC - Stiffness Score
Description: as for outcome 7
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 24
Percentage change | -35 (50.4)

9. Secondary Outcome: Change in WOMAC - Stiffness Score
Description: as for outcome 7
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 21
Percentage change | -43.30 (45.3)

10. Secondary Outcome: Change in WOMAC - Physical Function Score
Description: The WOMAC - Physical Function Score is calculated using the KOOS extension to the WOMAC score. The Physical Function Score comprises 17 items related to function in daily life and in sports/recreation; all items are rated on a Likert scale from 0-4; the total score is the sum of responses and ranges from 0-68. Higher scores indicate more severe dehabilitation.
Time Frame: Baseline, Month 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Percentage change | -51.20 (32.5)

11. Secondary Outcome: Change in WOMAC - Physical Function Score
Description: as for outcome 10
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 24
Percentage change | -47.8 (47.8)

12. Secondary Outcome: Change in WOMAC - Physical Function Score
Description: as for outcome 10
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 21
Percentage change | -49.90 (35.4)

13. Secondary Outcome: Change in WOMAC - Overall Score
Description: The WOMAC questionnaire includes 24 questions on daily activities. All items are rated on a scale from 0-4. The total score is the sum of responses and ranges from 0-96. A higher overall WOMAC score indicates greater pain, stiffness, and functional limitations.
Time Frame: Baseline, Month 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Percentage change | -47.50 (32.3)

14. Secondary Outcome: Change in WOMAC - Overall Score
Description: as for outcome 13
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 24
Percentage change | -48 (34.5)

15. Secondary Outcome: Change in WOMAC - Overall Score
Description: as for outcome 13
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 21
Percentage change | -48.10 (35.5)

16. Secondary Outcome: Change in Quality of Life Assessed Via 5-level EQ-5D Version (EQ-5D-5L)
Description: Quality of life reported by the patient measured using the 6-item EQ-5D-5L measure. EQ-5D-5L states are converted into an index value; index values range from full health (1) to no health (-0.109).
Time Frame: Baseline, Month 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 25
Percentage change | 19.80 (24.8)

17. Secondary Outcome: Change in Quality of Life Assessed Via EQ-5D-5L
Description: as for outcome 16
Time Frame: Baseline, Month 3
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 24
Percentage change | 17.6 (21)

18. Secondary Outcome: Change in Quality of Life Assessed Via EQ-5D-5L
Description: as for outcome 16
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | Embolization Group
Number analyzed (Participants) | 21
Percentage change | 20.6 (20)

ADVERSE EVENTS:
Time Frame: 12 months
Description: Study investigators monitor and screen for AEs at each visit.
Arm/Group | Embolization Group
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 11/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Embolization Group (N=25)
Skin discoloration (Skin and subcutaneous tissue disorders) | 4
Bone osteonecrosis (Musculoskeletal and connective tissue disorders) | 2
Burning sensation (Nervous system disorders) | 1
Access site hematoma / bruise (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/00/NCT04379700/Prot_SAP_001.pdf